CLINICAL TRIAL: NCT04601298
Title: The Risk Stratification of Papillary Thyroid Cancer With Bethesda Category III（AUS/FLUS）by Thyroid Fine-Needle Aspiration（FNA）Could be Assisted by Tumor Size for Precision Treatment
Brief Title: The Risk Stratification of Papillary Thyroid Cancer With AUS/FLUS by FNA
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Shen Qu, PI, Shanghai 10th People's Hospital
Other Study IDs: Bethesda Category III
Record Dates: First submitted 2020-09-29; First posted 2020-10-23 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Thyroid Cancer; Atypia of Undetermined Significance; FLUS
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AUS
- FLUS

INTERVENTIONS:
Other:

SUMMARY:
Purpose: To investigate the clinical characteristics of papillary thyroid cancer (PTC) with Bethesda category III (AUS/FLUS) by fine needle aspiration (FNA) and to assisted the precision treatment.

Methods:A total of 290 patients who underwent thyroidectomies or thyroid lobectomies from August 2015 to September 2020, following a diagnosis of Bethesda category III (AUS/FLUS) from preoperative thyroid FNA were investigated.

Groups: In order to investigate the clinopathologic characteristics, the patients, were grouped according to Cytology,Gender, Tumor size.

DETAILED DESCRIPTION:
Purpose: To investigate the clinical characteristics of papillary thyroid cancer (PTC) with Bethesda category III (AUS/FLUS) by fine needle aspiration (FNA) and to assisted the precision treatment.

Methods:A total of 1739 cases diagnosed with Bethesda category III (AUS/FLUS) by FNA from August 2015 to September 2020 were reviewed, and 523 patients received thyroidectomy or lobectomy. 290 patients were diagnosed with PTC and investigated retrospectively.

Groups: In order to investigate the clinopathologic characteristics, the patients, were grouped according to Cytology,Gender, Tumor size.as follows:AUS and FLUS&AUS/FLUS;male and female; tumor size≤1cm and>1cm.

ELIGIBILITY:
Inclusion Criteria:

Clinical cytology diagnosis of Bethesda category III (AUS/FLUS) pathological confirmation of thyroid malignancy after surgery.

Exclusion Criteria:

1. pathological confirmation of other thyroid carcinomas, including follicular carcinoma ,medullary carcinoma ,undifferentiated Spindle cell carcinoma and lymphoma were excluded
2. female who were pregnant were excluded
3. patients with mental disorders were excluded
4. patients without the complete clinical data were excluded

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The clinical database for patients undergoing thyroidectomies or thyroid lobectomies at the university hospital from August 2015 to September 2020 was revisited, and the thyroid pathology reports were screened and reviewed to analyse the comparison analysis of thyroid cancer with Bethesda category III (AUS/FLUS) by fine-needle aspiration cytology.
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Extra-thyroid extension | from 2015 to 2020
  Whether there is extension of the primary tumor outside of the thyroid capsule and invasion into surrounding structures. Analyze the correlation between extrathyroid infiltration and tumor size.

SECONDARY OUTCOMES:
Multifocality | from 2015 to 2020
  thyroid cancer lesions is more than two;analyze the correlation between multifocality and tumor size.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10Th People'S Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No